CLINICAL TRIAL: NCT06423677
Title: Evaluation of the Analgesic Efficacy of Serratus Posterior Superior Intercostal Plane (SPSIP) Block in Shoulder Arthroscopies: A Randomized Controlled Prospective Multicenter Study
Brief Title: Analgesic Efficacy of Serratus Posterior Superior Intercostal Plane (SPSIP) Block in Shoulder Arthroscopies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, Specialist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Serratus Posterior Superior
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative; Shoulder Pain; Block
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Bites and Stings | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- serratus posterior superior intercostal plane block + intravenous patient controlled analgesia (Active Comparator): serratus posterior superior intercostal plane block will be administered to these group. after the extubation intravenous patient controlled analgesia (PCA) will also be administered to patients.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block; Device: patient controlled analgesia
- intravenous patient controlled analgesia (Active Comparator): After the extubation, only intravenous patient controlled analgesia (PCA) will be administered to patients.
  Interventions: Device: patient controlled analgesia

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block — The Serratus Posterior Superior Intercostal Plane Block will be performed under ultrasound guidance. During the block, a linear ultrasound probe will be placed parallel to the spine of the scapula on the surgical side and then slid medially. The block needle will be advanced under ultrasound guidance over the 3rd rib. After the needle touches the rib, it will be withdrawn by 1mm, and the block site will be confirmed by injecting sterile 0.9% NaCl. Subsequently, patients will be administered 50mg of bupivacaine and 100mg of lidocaine in a controlled manner.
  Arms: serratus posterior superior intercostal plane block + intravenous patient controlled analgesia
Device: patient controlled analgesia — intravenous patient-controlled analgesia (PCA) with 4mg/ml Tramadol HCl in 100ml NaCl. There will be no basal infusion, with bolus doses of 20mg and a lockout period of 20 minutes, and a total dose limitation of 200mg over 4 hours

SUMMARY:
Patients in the block group will be placed in a lateral position with the operated shoulder on top before awakening from surgery. After ensuring aseptic conditions (the block site will be wiped three times with 10% povidone-iodine), the linear ultrasound probe will be covered in a sterile manner. While performing the block, the Hitachi brand linear ultrasound probe will be placed parallel to the scapular spine on the surgical side and will be slid medially. After imaging the 2nd and 3rd ribs on the medial side of the scapular spine, the block needle will be advanced under ultrasound guidance onto the 3rd rib. After contacting the rib with the needle, it will be retracted by 1mm, and the block site will be confirmed by injecting sterile 0.9% NaCl. Subsequently, patients will be administered 30ml of 0.25% bupivacaine in a controlled manner.

Before awakening, both the block group and the non-block group will be administered 1g of paracetamol and 1mg/kg of tramadol intravenously. In the postoperative period, these patients will be provided with multimodal analgesia, including intravenous patient-controlled analgesia (PCA) with 4mg/ml Tramadol HCl in 100ml NaCl. There will be no basal infusion, with bolus doses of 20mg and a lockout period of 20 minutes, and a total dose limitation of 200mg over 4 hours. Patients will be visited at 0, 1, 6, 12, and 24 hours, and they will be asked to draw their visual analog scale (VAS) score on a paper scale. The amount of opioid used in the PCA and the need for rescue analgesia (Arveles 50mg intravenously) will be assessed. Patients will routinely receive 4x1g paracetamol in the postoperative period.

DETAILED DESCRIPTION:
Patient Positioning and Preparation:

Patient Positioning:

Patients in the block group will be placed in a lateral position with the operated shoulder on top before awakening from surgery. This positioning facilitates access to the block site and ensures patient comfort.

Aseptic Technique:

The block site will be prepared by wiping it three times with 10% povidone-iodine to ensure asepsis.

The linear ultrasound probe will be covered in a sterile manner to prevent contamination during the procedure.

Ultrasound-Guided Block Procedure:

Probe Placement and Rib Identification:

The Hitachi brand linear ultrasound probe will be placed parallel to the scapular spine on the surgical side.

The probe will be slid medially to identify the 2nd and 3rd ribs on the medial side of the scapular spine. Accurate identification of these ribs is crucial for proper needle placement.

Needle Insertion and Block Site Confirmation:

A block needle will be advanced under ultrasound guidance onto the 3rd rib. The ultrasound guidance ensures precise needle placement, minimizing the risk of complications.

Once the needle contacts the rib, it will be retracted by 1mm. This slight retraction helps position the needle tip correctly for optimal drug delivery.

The block site will be confirmed by injecting sterile 0.9% NaCl. The spread of saline under ultrasound visualization confirms the correct location.

Anesthetic Administration:

Following confirmation of the block site, 30ml of 0.25% bupivacaine will be administered in a controlled manner. The controlled administration ensures a steady and effective distribution of the anesthetic agent.

Perioperative Analgesia Management:

Pre-Awakening Medication:

Before awakening from surgery, both the block group and the non-block group will receive:

1g of paracetamol intravenously.

1mg/kg of tramadol intravenously.

Postoperative Analgesia:

Postoperative analgesia will be managed using a multimodal approach, including:

Intravenous patient-controlled analgesia (PCA) with 4mg/ml Tramadol HCl in 100ml NaCl.

The PCA will be set with no basal infusion, allowing patients to self-administer bolus doses of 20mg with a lockout period of 20 minutes.

The total dose limitation will be set at 200mg over 4 hours to prevent overdose and manage pain effectively.

Postoperative Assessment and Follow-Up:

VAS Score Monitoring:

Patients will be visited at the following time intervals postoperatively: 0, 1, 6, 12, and 24 hours.

During each visit, patients will be asked to record their pain levels using the visual analog scale (VAS) on a paper scale. This subjective measure provides valuable insight into the patient's pain experience.

Opioid Consumption and Rescue Analgesia:

The amount of opioid used via PCA will be recorded to evaluate opioid consumption.

The need for rescue analgesia will be assessed and documented. If required, patients will receive 50mg of Arveles intravenously.

Routine Postoperative Medication:

All patients will receive routine postoperative medication, including 4x1g paracetamol to maintain baseline analgesia and reduce overall opioid requirements.

Randomization Process:

Randomization Protocol:

Patients scheduled for surgery will be randomly assigned to either the block group or the non-block group to ensure unbiased allocation and comparability between groups.

Randomization will be performed using a computer-generated random number sequence, ensuring that each patient has an equal chance of being allocated to either group.

Allocation concealment will be maintained by using opaque, sealed envelopes containing the group assignments. These envelopes will only be opened after patient consent and immediately before the block procedure.

Blinding:

The study will implement a single-blind design where the patients will be unaware of their group assignment to minimize bias in self-reported outcomes.

The healthcare providers responsible for postoperative care and outcome assessment will also be blinded to the group allocation to ensure objective evaluation of the study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining consent from the patient and their relative
* ASA score of I-II
* No bleeding diathesis
* No history of anticoagulant use
* No history of neuropathic diseases such as Diabetes Mellitus
* Patients aged 18-65 years undergoing shoulder arthroscopy surgery

Exclusion Criteria:

* Lack of consent from the patient or their relative
* Patients with an ASA score of III or above
* Patients with a history of bleeding diathesis
* Conditions where regional anesthesia is contraindicated
* Patients with a history of neuropathic diseases
* Patients under 18 years or over 65 years of age
* Patients with a history of allergies to the aforementioned medications
* Patients with an infection at the site where the block will be administered

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale score | 0, 1, 6, 12, and 24 hours
  Patients will be visited at 0, 1, 6, 12, and 24 hours, and they will be asked to draw their visual analog scale (VAS) score on a paper scale.0 means no pain, 10 means the most intense pain. 4 or more Visual analog scale scores means patients need rescue analgesia.
opioid consumption | 0, 1, 6, 12, and 24 hours
  Patients will be visited at 0, 1, 6, 12, and 24 hours and opioid consumption in the patient controlled analgesia device will be noted.0 means no pain, 10 means the most intense pain. 4 or more Visual analog scale scores means patients need rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)